CLINICAL TRIAL: NCT01453374
Title: A Phase 4, Pilot, Open-label Study of VIVITROL in the Prevention of Re-arrest and Re-incarceration
Brief Title: A Study of VIVITROL in the Prevention of Re-arrest and Re-incarceration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK21-028
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; VIVITROL; criminal justice
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIVITROL (Experimental): 380 mg IM injection
  Interventions: Drug: VIVITROL 380mg

INTERVENTIONS:
Drug: VIVITROL 380mg — 380 mg IM injection given once monthly

SUMMARY:
This phase 4 study will evaluate the feasibility of initiating subjects on VIVITROL in prison and continuing VIVITROL upon release into the community.

DETAILED DESCRIPTION:
This is an open-label study with a pre-post design. Pre-release opioid-dependent subjects from 4 Baltimore, MD area prisons (three for men and one for women) will receive 1 injection of VIVITROL prior to release from prison and will be offered 6 monthly injections of VIVITROL for 6 months post release. Subjects will complete follow-up visits 1 and 2 months after the last VIVITROL injection. Subjects will be assessed at 10 time points, and adherence to VIVITROL, both in prison and in the community, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Not currently addicted to opioids, but has a diagnosis of pre-incarceration opioid dependence
* Inmate at the Metropolitan Transition Center (Baltimore, MD), Maryland Correctional Institute for Women (Jessup, MD), Baltimore Pre-Release Unit (Baltimore, MD), or Jessup Pre-Release Unit (Jessup, MD) and eligible for release within 30 days of screening
* Expressing a goal of opiate-free treatment upon release
* Currently opioid free
* Planning to live in the Baltimore, MD area for at least 8 months following prison release

Exclusion Criteria:

* Pregnancy and/or breastfeeding
* Clinically significant active medical condition
* Active hepatitis
* Past or present history of an AIDS-indicator disease in subjects who are infected with HIV
* Any untreated or unstable psychiatric disorder(eg, bipolar with mania)
* Recent suicidal ideation
* Current chronic pain diagnosis for which opioids are prescribed
* Positive drug test for opioids
* History of drug overdose within the past 3 years requiring inpatient hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L Silverman, MD, Study Director — Alkermes, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-release opioid-dependent subjects from 4 Baltimore, MD area prisons (3 for men and 1 for women) received 1 injection of VIVITROL prior to release from prison and were offered 6 monthly injections of VIVITROL after release from prison, for a total of 7 injections.
Pre-assignment Details: Eligible subjects had a diagnosis of opioid dependence, were seeking treatment, and were eligible for release from prison within 30 days from screening.
Period: Overall Study
Arm/Group | VIVITROL
Started | 27
Completed | 9 (Defined as receiving 7 injections and 2 follow-up visits.)
Not Completed | 18
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5
Not completed — Incarcerated | 2

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 injection of VIVITROL
Arm/Group | VIVITROL
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Subject Re-arrest
Description: Subjects were considered to have had a re-arrest for any new crime or probation/parole violation if the subject had re-arrest records in the official criminal justice records and/or via self-report.
Time Frame: 7 months
Population: All subjects with non-missing data who received at least 1 injection of VIVITROL; 1 subject did not have any outcome data
Measure: Number; unit: participants re-arrested
Groups:
- <7 Injections: Subjects who received less than 7 VIVITROL injections
- All 7 Injections: Subjects who received all 7 VIVITROL injections
Arm/Group | <7 Injections | All 7 Injections
Number analyzed (Participants) | 16 | 10
participants re-arrested | 6 | 2
Statistical Analysis 1: Comparison: <7 Injections vs All 7 Injections; Test type: Superiority or Other; p > 0.05, Fisher Exact

2. Secondary Outcome: Incidence of Subject Re-incarceration
Description: Subjects were considered to have had a re-incarceration, a sentence to jail and/or prison, if the subject had re-incarceration records in the official criminal justice records and/or via self-report.
Time Frame: 7 months
Population: as for outcome 1
Measure: Number; unit: participants re-incarcerated
Arm/Group | <7 Injections | All 7 Injections
Number analyzed (Participants) | 16 | 10
participants re-incarcerated | 5 | 2
Statistical Analysis 1: Comparison: <7 Injections vs All 7 Injections; Test type: Superiority or Other; p > 0.05, Fisher Exact

3. Secondary Outcome: Opioid Use
Description: Opioid use was obtained via self-report on the Addiction Severity Index (ASI) or via a urine drug test.
Time Frame: 7 months
Population: All subjects with non-missing data who had at least 1 injection of VIVITROL; 1 subject did not have any outcome data
Measure: Number; unit: participants with positive opioid use
Arm/Group | <7 Injections | All 7 Injections
Number analyzed (Participants) | 16 | 10
participants with positive opioid use | 11 | 2
Statistical Analysis 1: Comparison: <7 Injections vs All 7 Injections; Test type: Superiority or Other; p < 0.05, Fisher Exact

4. Secondary Outcome: Opioid Overdose
Description: Number of subjects who overdosed during the study; measured through reported AEs of "overdose" and Opiate Overdose Form. The Form asks subjects if subjects overdosed during the past 30 days and, if so, how many times.
Time Frame: 7 months
Population: All subjects who received at least 1 injection of VIVITROL
Measure: Number; unit: participants who overdosed
Arm/Group | VIVITROL
Number analyzed (Participants) | 27
participants who overdosed | 1

5. Secondary Outcome: Drug Abuse Treatment Program Entry
Description: Number of subjects who participated in a drug treatment program during the study; assessed by review of Treatment Services Form.
Time Frame: 7 months
Population: as for outcome 1
Measure: Number; unit: participants who entered drug treatment
Arm/Group | VIVITROL
Number analyzed (Participants) | 26
participants who entered drug treatment | 24

6. Secondary Outcome: Retention in the Community
Description: Number of subjects who received all 6 post-release VIVITROL injections
Time Frame: 6 months
Population: All subjects who received at least 1 injection of VIVITROL
Measure: Number; unit: participants received all 7 injections
Arm/Group | VIVITROL
Number analyzed (Participants) | 27
participants received all 7 injections | 10

7. Secondary Outcome: Opioid Craving
Description: Change from baseline in peak craving score 30 days post last injection; assessed using a 100 mm visual analog scale (VAS). Subjects are asked to make 1 slash mark through a point on a 100 mm line that best describes their greatest craving for opioids, whereby 0 represents no craving and 100 is more than ever.
Time Frame: 8 months
Population: All subjects with non-missing data who received at least 1 injection of VIVITROL
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VIVITROL
Number analyzed (Participants) | 24
units on a scale
  Actual Value | 21.0 (33.4)
  Change from Baseline | -11.0 (47.4)

8. Secondary Outcome: Opioid Dependence
Description: Meeting Diagnostic Statistical Manual, version IV, text revision (DSM-IV-TR) criteria for opioid dependence
Time Frame: 7 months
Reporting Status: Not Posted

9. Secondary Outcome: Cocaine Use
Description: Number of subjects who used cocaine during the study; assessed using the Addiction Severity Index (ASI) and urine drug tests
Time Frame: 6 months
Population: All subjects with non-missing data who received at least 1 injection of VIVITROL
Measure: Number; unit: participants who used cocaine
Arm/Group | <7 Injections | All 7 Injections
Number analyzed (Participants) | 13 | 9
participants who used cocaine | 5 | 0
Statistical Analysis 1: Comparison: <7 Injections vs All 7 Injections; Test type: Superiority or Other; p < 0.10, Fisher Exact

10. Secondary Outcome: Criminal Activity
Description: Number of subjects who conducted any criminal activity during the study; assessed by review of criminal justice records and completion of the ASI and supplemental questionnaires
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants with criminal activity
Arm/Group | VIVITROL
Number analyzed (Participants) | 26
participants with criminal activity | 18

ADVERSE EVENTS:
Time Frame: Data were collected during a 9-month time frame
Arm/Group | VIVITROL
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIVITROL (N=27)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIVITROL (N=27)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Oedema peripheral (General disorders) | 4 (4)
Chest pain (General disorders) | 3 (6)
Injection site nodule (General disorders) | 2 (3)
Pain (General disorders) | 2 (3)
Injection site pain (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Blood glucose increased (Investigations) | 5 (5)
Platelet count increased (Investigations) | 5 (5)
Urine analysis abnormal (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3)
CSF specific gravity increased (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 3 (3)
Urine ketone body present (Investigations) | 3 (3)
Weight decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 3 (3)
Haematocrit decreased (Investigations) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (6)
Dizziness (Nervous system disorders) | 3 (3)
Depression (Psychiatric disorders) | 8 (10)
Anxiety (Psychiatric disorders) | 4 (4)
Stress (Psychiatric disorders) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2)
Drug withdrawal syndrome (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 11 (13)

LIMITATIONS AND CAVEATS:
The outcome measure of opioid dependence was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of such disclosure must be given to Alkermes for review at least 60 days prior to submission for publication. Revision to such disclosure will be negotiated in good faith by the Institution, Principal Investigator, and Alkermes. The disclosure may be submitted for publication or presented by the Institution and Principal Investigator only following receipt of written notice from an authorized representative of Alkermes stating that the disclosure has been reviewed and approved.